CLINICAL TRIAL: NCT03847909
Title: A Phase 2 Placebo-Controlled, Double-Blind, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of DCR-PHXC Solution for Injection (Subcutaneous Use) in Patients With Primary Hyperoxaluria
Brief Title: A Study to Evaluate DCR-PHXC in Children and Adults With Primary Hyperoxaluria Type 1 and Primary Hyperoxaluria Type 2
Acronym: PHYOX2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCR-PHXC-201
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Primary Hyperoxaluria Type 1 (PH1); Primary Hyperoxaluria Type 2 (PH2); Kidney Diseases; Urologic Diseases; Genetic Disease
Keywords: PH1; PH2; Primary Hyperoxaluria; RNAi; RNAi therapeutic; GalNAc; LDHA gene; LDH; siRNA
MeSH Terms: conditions — Primary hyperoxaluria type 1; Primary hyperoxaluria type 2; Kidney Diseases; Urologic Diseases; Genetic Diseases, Inborn; Hyperoxaluria, Primary | interventions — nedosiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DCR-PHXC (Experimental): Intervention, drug, DCR-PHXC
  Interventions: Drug: DCR-PHXC
- Placebo - Sterile Normal Saline (0.9% NaCl) (Placebo Comparator): Placebo, sterile normal saline (0.9% NaCl) for subcutaneous (SC) injection
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: DCR-PHXC — Multiple fixed doses of DCR-PHXC by subcutaneous (SC) injection
  Other Names: nedosiran
  Arms: DCR-PHXC
Drug: Sterile Normal Saline (0.9% NaCl) — Sterile Normal Saline (0.9% NaCl) for subcutaneous (SC) injection, administered at same injection volume as DCR-PHXC, to serve as placebo
  Arms: Placebo - Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of DCR-PHXC in Children and Adults with Primary Hyperoxaluria Type 1 (PH1) and Primary Hyperoxaluria Type 2 (PH2)

ELIGIBILITY:
Key Inclusion Criteria:

* Capable and willing to provide written informed consent or assent
* Documented diagnosis of PH1 or PH2, confirmed by genotyping
* Must meet the 24 hour urine oxalate excretion requirements
* Less than 20% variation between the two 24-hour urinary creatinine excretion values derived from the two 24-hour urine collections in the screening period
* Estimated GFR at screening ≥ 30 mL/min normalized to 1.73 m2 BSA

Key Exclusion Criteria:

* Renal or hepatic transplantation (prior or planned within the study period)
* Currently on dialysis or anticipated requirement for dialysis during the study period
* Plasma oxalate >30 µmol/L
* Documented evidence of clinical manifestations of systemic oxalosis (including pre-existing retinal, heart, or skin calcifications, or history of severe bone pain, pathological fractures, or bone deformations)
* Use of an RNA interference (RNAi) drug within the last 6 months
* Participation in any clinical study in which you received an investigational medicinal product (IMP) within 4 months before Screening
* Liver function test (LFT) abnormalities: Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 times upper limit of normal (ULN) for age and gender
* Inability or unwillingness to comply with study procedures

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (26):
- United States (5):
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Pittsburgh, Pennsylvania
- Australia (2):
  - Clinical Trial Site, Herston
  - Clinical Trial Site, Parkville
- Clinical Trial Site, Hamilton, Canada
- France (2):
  - Clinical Trial Site, Bron
  - Clinical Trial Site, Paris
- Germany (2):
  - Clinical Trial Site, Bonn
  - Clinical Trial Site, Heidelberg
- Clinical Trial Site, Jerusalem, Israel
- Clinical Trial Site, Roma, Italy
- Japan (3):
  - Clinical Trial Site, Nagoya
  - Clinical Trial Site, Tochigi
  - Clinical Trial Site, Tokyo
- Clinical Trial Site, Beirut, Lebanon
- Clinical Trial Site, Amsterdam, Netherlands
- Clinical Trial Site, Auckland, New Zealand
- Clinical Trial Site, Bialystok, Poland
- Clinical Trial Site, Bucharest, Romania
- Spain (2):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Santa Cruz
- United Kingdom (2):
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, Gamallo P, Rawson V. Population Pharmacokinetic and Pharmacodynamic Modelling and Simulation for Nedosiran Clinical Development and Dose Guidance in Pediatric Patients with Primary Hyperoxaluria Type 1. Clin Pharmacokinet. 2025 Sep;64(9):1395-1411. doi: 10.1007/s40262-025-01540-1. Epub 2025 Jul 2. PMID 40601241
- [Derived] Cox JH, Boily MO, Caron A, Sheng T, Wu J, Ding J, Gaudreault S, Chong O, Surendradoss J, Gomez R, Lester J, Dumais V, Li X, Gumpena R, Hall MD, Waterson AG, Stott G, Flint AJ, Moore WJ, Lowther WT, Knight J, Percival MD, Tong V, Oballa R, Powell DA, King AJ. Characterization of CHK-336, A First-in-Class, Liver-Targeted, Small-Molecule Lactate Dehydrogenase Inhibitor for Hyperoxaluria Treatment. J Am Soc Nephrol. 2025 Apr 7;36(8):1535-1547. doi: 10.1681/ASN.0000000690. PMID 40193200
- [Derived] Baum MA, Langman C, Cochat P, Lieske JC, Moochhala SH, Hamamoto S, Satoh H, Mourani C, Ariceta G, Torres A, Wolley M, Belostotsky V, Forbes TA, Groothoff J, Hayes W, Tonshoff B, Takayama T, Rosskamp R, Russell K, Zhou J, Amrite A, Hoppe B; PHYOX2 study investigators. PHYOX2: a pivotal randomized study of nedosiran in primary hyperoxaluria type 1 or 2. Kidney Int. 2023 Jan;103(1):207-217. doi: 10.1016/j.kint.2022.07.025. Epub 2022 Aug 22. PMID 36007597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 sites in France, Spain, Italy, Netherlands, Germany, United Kingdom, Australia, United States, Canada, Lebanon, and Japan.
Pre-assignment Details: A total of 57 participants were screened, of which 35 participants were randomized: 23 to DCR-PHXC and 12 to placebo. All 35 randomized participants received at least one dose of study drug.
Groups:
- DCR-PHXC: Participants aged greater than or equal to (>=) 12 years weighing >=50 kilograms (kg) received nedosiran 170 milligram (mg) (160 milligrams per millilitre [mg/mL] free acid equivalent [FAE]); participants >=12 years weighing less than (<) 50 kg received 136 mg (128 mg FAE); and participants 6-11 years received 3.5 milligrams per kilogram (mg/kg) (3.3 mg/kg FAE) not exceeding 136 mg, subcutaneous (SC) injection into the abdomen or thigh on Days 1, 30, 60, 90, 120 and 150.
- Placebo: Participants received the equivalent volume of nedosiran matching placebo SC injection into the abdomen or thigh on Days 1, 30, 60, 90, 120 and 150.
Period: Overall Study
Arm/Group | DCR-PHXC | Placebo
Started | 23 | 12
Safety Population | 23 | 12
Intent to Treat (ITT) Population | 23 | 12
Modified ITT (MITT) Population | 22 | 12
Completed | 22 | 11
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- DCR-PHXC: Participants aged >=12 years weighing >=50 kg received nedosiran 170 mg (160 mg/mL FAE); participants >=12 years weighing <50 kg received 136 mg (128 mg FAE); and participants 6-11 years received 3.5 mg/kg (3.3 mg/kg FAE) not exceeding 136 mg, SC injection into the abdomen or thigh on Days 1, 30, 60, 90, 120 and 150.
- Total: Total of all reporting groups
Arm/Group | DCR-PHXC | Placebo | Total
Number analyzed (Participants) | 23 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (11.95) | 23.6 (11.48) | 23.7 (11.62)
Age, Customized [Count of Participants; unit: Participants]
  Between 2 to 11 years | 3 | 2 | 5
  Between 12 to 17 years | 6 | 4 | 10
  Between 18 to 64 years | 14 | 6 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 19 | 11 | 30
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 10 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: AUC From Day 90 To Day 180, Based on Percent Change From Baseline in 24-Hour Uox
Description: The AUC of 24-hour urinary oxalate (Uox) from Day 90 to Day 180, based on percent change from baseline, was compared between the active treatment group and placebo group. A multiple imputation approach was used to handle missing Uox data and then calculate the AUC.
Time Frame: From Day 90 to 180
Population: MITT population included all participants in the ITT population who had at least one efficacy assessment after the Day 90 dosing visit, where the ITT population included all participants who were randomized and had at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Percent change in 24-hour Uox AUC
Groups:
- DCR-PHXC: Participants aged >=12 years weighing >=50 kg received nedosiran 170 mg (160 mg/mL FAE); participants >=12 years weighing <50 kg received 136 mg (128 mg FAE); and participants 6-11 years received 3.5 mg/kg (3.3 mg/kg free acid equivalent [FAE]) not exceeding 136 mg, SC injection into the abdomen or thigh on Days 1, 30, 60, 90, 120 and 150.
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 12
Percent change in 24-hour Uox AUC | 3507.4 (788.49) | -1664.4 (1189.96)
Statistical Analysis 1: Comparison: DCR-PHXC vs Placebo; Test type: Superiority — P value is from an ANCOVA model with treatment group as the main effect, age category, baseline eGFR category, baseline Uox value as covariates for adjustment; p < 0.0001, ANCOVA; Difference of Least Mean Square = 5171.7, 95% CI 2-sided [2929.3 to 7414.2], Standard Error of Mean 1144.07

2. Secondary Outcome: Percentage of Participants Whose 24-hour Uox Values Normalized or Near-normalized on at Least 2 Consecutive Visits
Description: Percentage of participants whose 24-hour Uox values normalized or near-normalized on at least 2 consecutive visits are presented. Normalization of Uox was defined as less than (<) 0.46 millimole per 24 hours (mmol/24 hours) and near normalization was defined as greater than or equal to (>=) 0.46 to < 0.60 mmol/24 hours (values adjusted per 1.73 square meter [1.73 m^2] body surface area [BSA] in participants aged <18 years).
Time Frame: From Day 90 to 180
Population: Modified Intent-to-treat population (MITT) included all participants in the intent-to-treat (ITT) population who had at least one efficacy assessment after the Day 90 dosing visit where ITT population included all participants who were randomized and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 12
Percentage of participants | 50 | 0

3. Secondary Outcome: Percent Change From Baseline to Day 180 in the Summed Surface Area of Kidney Stones
Description: Percent change from baseline to Day 180 in the summed surface area measured in millimetre square (mm^2) of kidney stones is presented.
Time Frame: Baseline, Day 180
Population: The ITT population included all participants who were randomised and had at least one post-baseline efficacy assessment. Number of participants analysed signifies participants with available data.
Measure: Median (Full Range); unit: Percent change in summed surface area
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 16 | 10
Percent change in summed surface area | -2.13 [-100.0 to 228.6] | 21.77 [-24.3 to 1500.0]

4. Secondary Outcome: Percent Change From Baseline to Day 180 in the Number of Kidney Stones
Description: Percent change from baseline to Day 180 in the number of kidney stones is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 3
Measure: Median (Full Range); unit: Percent change in kidney stone numbers
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 16 | 10
Percent change in kidney stone numbers | 0.00 [-100.0 to 200.0] | 0.00 [-94.1 to 100.0]

5. Secondary Outcome: Percent Change From Baseline to Day 180 in Plasma Oxalate (For Adults Only)
Description: Percent change from baseline to Day 180 in plasma oxalate (for adults only) is presented.
Time Frame: Baseline, Day 180
Population: Analysis population included all adult participants from ITT population who were randomised and had at least one post-baseline efficacy assessment. Number of participants analysed signifies participants with available data.
Measure: Median (Full Range); unit: Percent change in plasma oxalate
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 14 | 5
Percent change in plasma oxalate | -25.00 [-61.9 to 22.2] | -0.00 [-25.0 to 350.0]

6. Secondary Outcome: Rate of Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline to Day 180
Description: Monthly rate of eGFR change is presented. eGFR was calculated using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) and creatinine-based equation.
Time Frame: Baseline, Day 180
Population: The ITT population included all participants who were randomised and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Error); unit: mL/minute/1.73 m^2
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 23 | 12
mL/minute/1.73 m^2 | 0.3533 (0.39610) | 1.1008 (0.54849)

7. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) And Serious Treatment Emergent Adverse Events (TEAEs)
Description: Number of TEAEs and TESAEs are presented. An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalisation, results in persistent disability/incapacity or is a congenital anomaly/birth defect. TEAE was defined as any AE with an onset date/time on or after administration (including any partial administration) of the first dose of study intervention and through the study completion date from the end of study case report form (CRF).
Time Frame: From Baseline up to Day 180
Population: The safety population included all participants randomly assigned to study intervention and who took at least 1 partial or full dose of study intervention.
Measure: Number; unit: Events
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 23 | 12
Events
  TEAEs | 101 | 54
  Serious TEAEs | 1 | 3

8. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG): Heart Rate
Description: Change from baseline in heart rate is presented.
Time Frame: Baseline, Day 180
Population: The safety population included all participants randomly assigned to study intervention and who took at least 1 partial or full dose of study intervention. Number of participants analysed signifies participants with available data.
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
beats per minute (beats/min) | 0.4 (8.36) | -1.8 (9.18)

9. Secondary Outcome: Change From Baseline in ECG: PR Interval, QRS Duration, QT Interval, QTcB Interval, QTcF Interval and RR Interval
Description: Change from baseline in PR interval, QRS duration, QT interval, QTcB interval, QTcF interval and RR interval is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
milliseconds (msec)
  PR interval | -0.5 (13.92) | 1.3 (8.14)
  QRS duration | 1.3 (6.01) | -1.5 (7.53)
  QT interval | -2.4 (23.73) | 4.0 (22.97)
  QTcB interval | -0.8 (15.60) | -0.7 (17.31)
  QTcF interval | -1.1 (15.80) | 1.2 (15.59)
  RR interval | -7.6 (99.35) | 17.8 (109.73)

10. Secondary Outcome: Number of Participants With Most Abnormal Post-Baseline Shift in Physical Examination
Description: Number of participants who had most abnormal post-baseline shift in physical examination are presented. Physical examination shifts were categories into 4 categories: 1) missing; 2) normal; 3) abnormal-not clinically significant (NCS) and 4) abnormal-clinically significant (CS). Each category was presented according body systems including: 1) eyes, ears, nose and throat; 2) chest/respiratory; 3) heart/cardiovascular; 4) gastrointestinal/liver; 5) musculoskeletal/extremities; 6) dermatological/skin; 7) thyroid/neck; 8) lymph nodes; 9) neurological.
Time Frame: Baseline up to Day 180
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 23 | 12
Participants
  Eyes, ears, nose and throat: missing | 1 | 1
  Eyes, ears, nose and throat: normal | 21 | 11
  Eyes, ears, nose and throat: abnormal-NCS | 1 | 0
  Eyes, ears, nose and throat: abnormal-CS | 0 | 0
  Chest/respiratory: missing | 0 | 0
  Chest/respiratory: normal | 23 | 12
  Chest/respiratory: abnormal-NCS | 0 | 0
  Chest/respiratory: abnormal-CS | 0 | 0
  Heart/cardiovascular: missing | 0 | 0
  Heart/cardiovascular: normal | 22 | 12
  Heart/cardiovascular: abnormal-NCS | 1 | 0
  Heart/cardiovascular: abnormal-CS | 0 | 0
  Gastrointestinal/liver: missing | 0 | 0
  Gastrointestinal/liver: normal | 22 | 8
  Gastrointestinal/liver: abnormal-NCS | 1 | 4
  Gastrointestinal/liver: abnormal-CS | 0 | 0
  Musculoskeletal/extremities: missing | 1 | 1
  Musculoskeletal/extremities: normal | 22 | 10
  Musculoskeletal/extremities: abnormal-NCS | 0 | 1
  Musculoskeletal/extremities: abnormal-CS | 0 | 0
  Dermatological/skin: missing | 0 | 0
  Dermatological/skin: normal | 18 | 8
  Dermatological/skin: abnormal-NCS | 4 | 4
  Dermatological/skin: abnormal-CS | 1 | 0
  Thyroid/neck: missing | 1 | 1
  Thyroid/neck: normal | 22 | 10
  Thyroid/neck: abnormal-NCS | 0 | 1
  Thyroid/neck: abnormal-CS | 0 | 0
  Lymph nodes: missing | 0 | 1
  Lymph nodes: normal | 23 | 10
  Lymph nodes: abnormal-NCS | 0 | 1
  Lymph nodes: abnormal-CS | 0 | 0

11. Secondary Outcome: Change From Baseline in Vital Signs: Height
Description: Change from baseline to Day 180 in height is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: centimetres (cm)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 11
centimetres (cm) | 0.70 (2.383) | 1.08 (1.446)

12. Secondary Outcome: Change From Baseline in Vital Signs: Weight
Description: Change from baseline to Day 180 in weight is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
kilograms | 1.134 (3.4794) | 1.350 (3.4330)

13. Secondary Outcome: Change From Baseline in Vital Signs: Body Mass Index (BMI)
Description: Change from baseline to Day 180 in BMI is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 11
Kilograms per square meter (kg/m^2) | 0.23 (1.175) | 0.14 (1.293)

14. Secondary Outcome: Change From Baseline in Vital Signs: Oral Body Temperature
Description: Change from baseline to Day 180 in oral body temperature is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Degree Celsius (C)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
Degree Celsius (C) | 0.01 (0.399) | 0.05 (0.446)

15. Secondary Outcome: Change From Baseline in Vital Signs: Heart Rate
Description: Change from baseline to Day 180 in heart rate is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
beats/minute | 0.8 (10.64) | -3.1 (6.35)

16. Secondary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: Change from baseline to Day 180 in respiratory rate is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 10
Breaths per minute | -0.2 (3.02) | -1.1 (5.00)

17. Secondary Outcome: Change From Baseline in Vital Signs: Systolic and Diastolic Blood Pressure
Description: Change from baseline to Day 180 in systolic and diastolic blood pressure is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
millimetres of mercury (mmHg)
  Systolic blood pressure | -2.0 (13.64) | -3.0 (9.82)
  Diastolic blood pressure | 0.8 (9.20) | -2.6 (11.84)

18. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Tests: Alanine Aminotransferase, Aspartate Aminotransferase, Glutamate Dehydrogenase, Gamma Glutamyl Transferase, Alkaline Phosphatase, Lactate Dehydrogenase and Creatine Kinase
Description: Change from baseline to Day 180 in alanine aminotransferase, aspartate aminotransferase, glutamate dehydrogenase, gamma glutamyl transferase, alkaline phosphatase, lactate dehydrogenase and creatine kinase are presented.
Time Frame: Baseline, Day 180
Population: The safety population included all participants randomly assigned to study intervention and who took at least 1 partial or full dose of study intervention. Number of participants analysed signifies participants with available data and number analysed signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Units per litre (U/L)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
Units per litre (U/L)
  Alanine aminotransferase | 1.0 (8.59) | -1.1 (4.59)
  Aspartate aminotransferase | -0.2 (4.95) | -1.3 (4.73)
  Glutamate dehydrogenase | -0.15 (1.913) | -0.38 (1.064)
  Gamma glutamyl transferase | 2.7 (4.12) | -0.2 (3.03)
  Alkaline phosphatase | 3.0 (29.11) | -16.8 (41.78)
  Lactate dehydrogenase: number analyzed (Participants) | 20 | 10
  Lactate dehydrogenase | 4.1 (20.51) | 1.0 (20.72)
  Creatine kinase | 7.5 (59.28) | -34.1 (160.46)

19. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Tests: Bilirubin, Direct Bilirubin and Creatinine
Description: Change from baseline to Day 180 in bilirubin, direct bilirubin and creatinine are presented.
Time Frame: Baseline, Day 180
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: micromoles per litre (umol/L)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
micromoles per litre (umol/L)
  Bilirubin | 1.0 (3.18) | 0.4 (1.80)
  Direct bilirubin: number analyzed (Participants) | 22 | 10
  Direct bilirubin | 0.1 (1.32) | 0.1 (0.32)
  Creatinine | -1.2 (10.81) | 4.3 (11.02)

20. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Tests: Protein, Albumin
Description: Change from baseline to Day 180 in protein and albumin are presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: grams per litre (g/L)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
grams per litre (g/L)
  Protein | 0.4 (4.47) | 1.5 (6.27)
  Albumin | 0.5 (3.22) | 1.2 (3.63)

21. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Tests: Sodium, Chloride, Potassium and Urea
Description: Change from baseline to Day 180 in sodium, chloride, potassium and urea are presented.
Time Frame: Baseline, Day 180
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/L)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 22 | 11
millimoles per litre (mmol/L)
  Sodium | 0.4 (2.44) | 0.2 (3.03)
  Chloride | 0.6 (3.30) | -0.4 (4.08)
  Potassium: number analyzed (Participants) | 21 | 10
  Potassium | -0.04 (0.425) | 0.05 (0.360)
  Urea | 0.01 (0.895) | 0.40 (1.197)

22. Secondary Outcome: Change From Baseline in Clinical Chemistry Laboratory Tests: Vitamin B6
Description: Change from baseline to Day 180 in vitamin B6 is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nanomoles per litre (nmol/L)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 2 | 3
nanomoles per litre (nmol/L) | 34.60 (99.278) | -215.73 (337.775)

23. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Erythrocytes
Description: Change from baseline to Day 180 in erythrocytes is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
10^12 cells per liter | -0.04 (0.365) | 0.02 (0.230)

24. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Hemoglobin and Erythrocytes Mean Corpuscular Hemoglobin Concentration
Description: Change from baseline to Day 180 in hemoglobin and erythrocytes mean corpuscular hemoglobin concentration are presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per litre (g/L)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
gram per litre (g/L)
  Hemoglobin | -1.7 (8.90) | 0.1 (6.62)
  Ery. mean corpuscular hemoglobin concentration | 1.5 (15.10) | -4.8 (10.80)

25. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Hematocrit
Description: Change from baseline to Day 180 in hematocrit is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Litre/litre (L/L)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
Litre/litre (L/L) | -0.004 (0.0271) | 0.006 (0.0288)

26. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Erythrocytes (Ery.) Mean Corpuscular Volume and Mean Platelet Volume
Description: Change from baseline to Day 180 in ery. mean corpuscular volume and mean platelet volume are presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
femtoliter (fL)
  Ery. mean corpuscular volume | 0.0 (2.31) | 1.1 (3.57)
  Mean platelet volume | -0.03 (0.864) | 0.61 (0.547)

27. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Erythrocytes Mean Corpuscular Hemoglobin
Description: Change from baseline to Day 180 in erythrocytes mean corpuscular hemoglobin is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: picogram (pg)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
picogram (pg) | -0.1 (1.37) | -0.1 (0.99)

28. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Reticulocytes, Platelets, Leukocytes, Lymphocytes, Monocytes, Eosinophils, Basophils, Neutrophils
Description: Change from baseline to Day 180 in reticulocytes, platelets, leukocytes, lymphocytes, monocytes, eosinophils, basophils, neutrophils are presented.
Time Frame: Baseline, Day 180
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
10^12 cells per liter
  Reticulocytes: number analyzed (Participants) | 20 | 9
  Reticulocytes | 0.2 (30.08) | -23.1 (32.21)
  Platelets | -11.4 (54.50) | 2.3 (53.30)
  Leukocytes | 0.18 (1.573) | -1.03 (1.931)
  Lymphocytes | -0.03 (0.621) | 0.06 (0.331)
  Monocytes | 0.07 (0.085) | -0.02 (0.103)
  Eosinophils | 0.03 (0.072) | 0.04 (0.126)
  Basophils | 0.01 (0.062) | -0.04 (0.097)
  Neutrophils | 0.14 (1.195) | -1.07 (1.700)

29. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Lymphocytes/Leukocytes
Description: Change from baseline to Day 180 in lymphocytes/leukocytes is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes/leukocytes
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
Percentage of lymphocytes/leukocytes | -1.3 (10.26) | 5.1 (10.21)

30. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Monocytes/Leukocytes
Description: Change from baseline to Day 180 in monocytes/leukocytes is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of monocytes/leukocytes
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
Percentage of monocytes/leukocytes | 1.0 (2.04) | 0.9 (2.51)

31. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Eosinophils/Leukocyte
Description: Change from baseline to Day 180 in eosinophils/leukocytes is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of eosinophils/leukocytes
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
Percentage of eosinophils/leukocytes | 0.4 (1.56) | 0.9 (1.66)

32. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Basophils/Leukocytes
Description: Change from baseline to Day 180 in basophils/leukocytes is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of basophils/leukocytes
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
Percentage of basophils/leukocytes | 0.0 (0.77) | 0.1 (0.74)

33. Secondary Outcome: Change From Baseline in Clinical Hematology Laboratory Tests: Neutrophils/Leukocytes
Description: Change from baseline to Day 180 in neutrophils/leukocytes is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils/leukocytes
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
Percentage of neutrophils/leukocytes | -0.3 (11.45) | -7.1 (13.14)

34. Secondary Outcome: Change From Baseline in Clinical Urinalysis Laboratory Tests: Specific Gravity
Description: Change from baseline to Day 180 in urine specific gravity is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per millilitre (g/mL)
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
gram per millilitre (g/mL) | 0.0000 (0.00872) | -0.0008 (0.00480)

35. Secondary Outcome: Change From Baseline in Clinical Urinalysis Laboratory Tests: pH
Description: Change from baseline to Day 180 in urine pH is presented.
Time Frame: Baseline, Day 180
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | DCR-PHXC | Placebo
Number analyzed (Participants) | 21 | 10
pH | 0.29 (1.067) | -0.10 (0.738)

36. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of DCR-PHXC
Description: The Cmax was defined as the maximum observed plasma concentration during a dosing interval. Data for this endpoint is reported only for adults and adolescent participants from PK population.
Time Frame: For adults: Day 1 and 30: predose, 5, 15, and 30 minutes and 1, 2, 4, 6, 10, and 12 hours (hrs) postdose; Day 150: predose, 2, 6, and 12 hours postdose For adolescents: Days 1 and 30: predose, 30 minutes and 2 and 10 hours postdose
Population: The Pharmacokinetic (PK) population included all participants in the safety population without major dosing violations, where safety population included all participants randomly assigned to study intervention and who took at least 1 partial or full dose of study intervention. Number of participants analysed signifies participants with available data and number analysed signifies participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Groups:
- DCR-PHXC: Adults: Participant analysis set included all adult participant (age >= 18 years) from DCR-PHXC arm who received 170 mg nedosiran.
- DCR-PHXC: Adolescents: Participants analysis set included all adolescents (aged 12-17 years) from DCR-PHXC arm who received 170 mg nedosiran.
Arm/Group | DCR-PHXC: Adults | DCR-PHXC: Adolescents
Number analyzed (Participants) | 12 | 5
nanogram per millilitre (ng/mL)
  Day 1 | 778 (35.7) | 363 (76.7)
  Day 30: number analyzed (Participants) | 11 | 5
  Day 30 | 774 (46.1) | 350 (48.6)
  Day 150: number analyzed (Participants) | 8 | 0
  Day 150 | 648 (55.5) |

37. Secondary Outcome: Area Under the Curve From Time of Administration to the Last Measurable Concentration (AUC0-last) of of DCR-PHXC
Description: AUC0-last was defined as the area under the curve from time of administration to the last measurable concentration. Data for this endpoint is reported only for adults and adolescent participants from PK population.
Time Frame: For adults: Day 1 and 30: predose, 5, 15, and 30 minutes and 1, 2, 4, 6, 10, and 12 hours postdose; Day 150: predose, 2, 6, and 12 hours postdose For adolescents: Days 1 and 30: predose, 30 minutes and 2 and 10 hours postdose
Population: The PK population included all participants in the safety population without major dosing violations, where safety population included all participants randomly assigned to study intervention and who took at least 1 partial or full dose of study intervention. Number of participants analysed signifies participants with available data and number analysed signifies participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per millilitre (h*ng/mL)
Arm/Group | DCR-PHXC: Adults | DCR-PHXC: Adolescents
Number analyzed (Participants) | 12 | 5
hours*nanograms per millilitre (h*ng/mL)
  Day 1 | 12500 (29.3) | 6450 (54.5)
  Day 30: number analyzed (Participants) | 11 | 5
  Day 30 | 12800 (38.4) | 6400 (45.1)
  Day 150: number analyzed (Participants) | 8 | 0
  Day 150 | 6100 (46.2) |

ADVERSE EVENTS:
Time Frame: From Day 1 up to end of the study (Day 180)
Description: The safety population included all participants randomly assigned to study intervention and who took at least 1 partial or full dose of study intervention. All serious and non-serious adverse events presented here are treatment emergent adverse events.
Arm/Group | DCR-PHXC | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/12
Other Adverse Events (participants affected / at risk) | 16/23 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DCR-PHXC (N=23) | Placebo (N=12)
Tachycardia (Cardiac disorders) | 1 | 0
Blood creatinine increased (Blood and lymphatic system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DCR-PHXC (N=23) | Placebo (N=12)
Injection site erythema (General disorders) | 5 | 0
Injection site pain (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Glutamate dehydrogenase increased (Investigations) | 0 | 1
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 4 | 3
Sensory disturbance (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Renal colic (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SPONSOR agrees that the Principal Investigator shall have the right to publish or permit the publication of any information or material relating to or arising out of the work after prior submittal to SPONSOR provided that if SPONSOR shall so request, the investigator will delay publication for a maximum of ninety (90) days after submittal to SPONSOR to enable SPONSOR to protect its rights. SPONSOR will comment on such documents within thirty (30) days.

DOCUMENTS (2):
  • Study Protocol (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT03847909/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT03847909/SAP_001.pdf